CLINICAL TRIAL: NCT05304624
Title: Comparison of Er,Cr:YSGG Laser and Diode Laser in the Treatment of Gingival Melanin Pigmentation: Randomised Clinical Trial
Brief Title: Comparison of Er,Cr:YSGG Laser and Diode Laser in the Treatment of Gingival Melanin Pigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Ekin Besiroglu, assistant profesor, Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-68869993-511
Record Dates: First submitted 2022-03-11; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Pigmentation
Keywords: Er,Cr:YSGG laser; Diode Laser; Gingival pigmentation
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: ErCr:YSGG laser (Active Comparator): Waterlase iPlus,Biolase-USA Er,Cr:YSGG laser (2780nm) was set at frequency 50Hz, power of 2.5W and 1562.5 W/cm2. MZ6 (400µm fiber tip) was used in contact mode for de-epitelization procedure.
  Another visit of laser ablation was performed after 7 days to remove the remaining pigmentation. The same laser settings were used.
  Interventions: Device: laser
- Group 2: Diode laser (Experimental): Ilase, Biolase-USA Diode laser (940nm) was set at power of 1.2W and 750 W/cm2. 400µm fiber tip was used in contact mode and continuous-wave for de-epitelization procedure.
  Another visit of laser ablation was performed after 7 days to remove the remaining pigmentation. The same laser settings were used.
  Interventions: Device: laser

INTERVENTIONS:
Device: laser — these lasers are routinely used in dental practice

SUMMARY:
The main aim of this paper is to explore the efficiancy on the extention and density of pigmentation between diode and Er,Cr:YSGG lasers. The second aim of this study was to investigate the lasers effects of patient pain and comfort.

DETAILED DESCRIPTION:
Recently, soft tissue aesthetics has become an important issue in dentistry. The normal physiological color of the gingiva is coral pink or pale pink. The color of gingiva is determined by several factors, including thickness of ephitelium, degree of keratinization, the number and size of underlying blood vessels and pigments within the epithelium. Gingival hyperpigmentation is caused by excessive deposition of melanin located in the basal and suprabasal cell layers of the epithelium. Many etiological factors such as smoking can stimulate melanin pigmentation. It has been reported that polycyclic amines such as nicotine and benzopyrene, which are known to penetrate melanocytes and bind to melanin, in cigarettes cause stimulation of melanocytes and as a result increase melanin production. Smoker melanocyte pigmentation was described first time by Hedin in 1977 as 'a local benign melanin pigmentation often seen in the attached gingiva'. Although physiologic melanin pigmentation and smoker melanosis are not medical problems, patients seek treatment for esthetic purposes. Various depigmentation techniques are employed to address the aesthetic concerns of individuals. Methods used for depigmentation: Chemical treatment, electrosurgery, abrasion with diamond tools, scalpel technique, gingivectomy, gingival graft, cryosurgery and lasers. Which method to choose depends on clinical experience and individual preferences. However, most researchers consider laser ablation to be more effective, convenient, and safer for gingival depigmentation. Many laser systems such as CO2 laser, Diyot laser, Neodymium Doped:Yttrium Aluminum Garnet(Nd:YAG) laser, Erbium Doped:Yttrium Aluminum Garnet(Er:YAG) laser and Erbium Chromium-Doped:Yttrium, Scandium, Gallium, Garnet(Er,Cr:YSGG) are used for this purpose. In melanin depigmentation with laser, the ability melanocytes which containing melanin to absorb the laser beam depends on the wavelength and water. The wavelength of the Er,Cr:YSGG laser is 2780nm, while the wavelength of the diode laser is 810-980nm.10 While diode laser is used for soft tissue surgery, Er,Cr:YSGG laser is used for soft and hard tissue surgery. Although there are more case reports regarding the use of diode lasers in gingival depigmentation, only a few focus on the use of Er, Cr:YSGG laser. In this study; in the treatment of gingival depigmentation by use of Er, Cr: YSGG laser and Diode laser to patients, it was aimed to evaluate the satisfaction of the patients during and after the operation, to evaluate the change in gingival tissue thickness and to evaluate the rate of repigmentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic healthy or not taking any medication
* Patients who are not pregnant or breastfeeding
* Patients between 18-40 years old
* Physiologic gingival hyperpigmentation on the facial aspect of maxillary first right premolar to first left premolar region
* Patients with esthetic concerns
* Patients who have smoked at least 10 cigarettes per day for at least 5 years
* Periodontally healthy patients

Exclusion Criteria:

* Patients with any systemic diseases or taking any medication
* Pregnant and lactating women
* Patients under 18 years
* Patients without gingival melanin pigmentation on the facial aspect of maxillary first right premolar to first left premolar region
* Patients who smoke less than 5 years and/or less than 10 cigarettes per day
* Non-smokers
* Patients with any metallic restoration or undergoing orthodontic treatment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
depigmentation with two different laser devices | 1 year
  Dummett Oral Pigmentasyon Indeks (DOPI) tehat identifies pigmentation as score 1- no clinical pigmentation (pink tissue), score 2-mild clinical pigmentation (light brown), score 3-moderate clinical pigmentation (mixed brown and pink), and score 4-heavy clinical pigmentation (deep brown to bluish black).
  Photographic Image Assesment: All photographs were taken in a standardized environment by using a Canon EOS 700D with Macro Lens EF 100 mm with automatic focusing. All photographs were taken at a standard distance which was 30 cm as recorded from the patient's cental teeth to the edge of the camera lens. The periodontal probe was used for the calibration of intraoral photographs. Photographs were analyzed with ImageJ Software version10.2. The pigmented areas on the photograph will be calculated in mm2.

SECONDARY OUTCOMES:
Pain Perception | 1 year
  The visual analog scale (VAS) was used at intraoperatively, 1st day and 1st week post-operative visits to measure the intensity of pain experienced during and after the treatment. The patients were asked to rate the degree of pain, on a 10 cm horizontal VAS by placing a vertical mark to assess position between the two end-points (from no-pain to severe-pain).
Patient Esthetic Satisfaction | 1 year
  Another VAS was used in the 12th month for evaluation of patient esthetic satisfaction. The patients were asked to rate the degree of esthetic satisfaction, on a 10 cm horizontal VAS by placing a vertical mark to assess position between the two end-points (from not at all to very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Ekin Beşiroğlu, Principal Investigator — Istanbul Okan University, Istanbul
Locations (1):
- Istanbul Okan University, Istanbul, Tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Besiroglu-Turgut E, Kayaalti-Yuksek S. Comparison of Er,Cr:YSGG laser and diode laser in the treatment of gingival melanin pigmentation: a randomized clinical trial. Lasers Med Sci. 2023 Feb 27;38(1):79. doi: 10.1007/s10103-023-03738-w. PMID 36847909